CLINICAL TRIAL: NCT04300725
Title: Video Counseling: A Randomized Control Trial Comparing Video Counseling and Verbal Counseling in Patients Undergoing an Induction of Labor.
Brief Title: Video Counseling: A Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Kevin Marques, Assistant Professor Department of Obstetrics, Gynecology and Women's Health, University of Louisville
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 19.0271
Record Dates: First submitted 2020-02-25; First posted 2020-03-09 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Pregnancy Related
Keywords: Induction of Labor; Video Counseling

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: • Randomization will occur after informed written consent has been obtained. Treatment randomization will be performed using a block randomization approach with block sizes of 10 individuals. A list will be created using www.sealedenvelope.com, and these will be placed in numbered envelopes to be opened after patient consent by the intern resident.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verbal Counseling (No Intervention): Patients in one study arm receive only verbal counseling prior to their induction of labor.
- Video Counseling (Experimental): Patients in other study arm will receive verbal + video counseling prior to their induction of labor.
  Interventions: Other: Video Counseling

INTERVENTIONS:
Other: Video Counseling — Patients in the other study arm receive verbal + video counseling prior to their induction of labor.
  Arms: Video Counseling

SUMMARY:
Lack of standardized verbal counseling prior to an induction of labor can leave many patients feeling uninformed and unprepared. The purpose of this blinded, randomized controlled trial was to compare video vs verbal counseling in a cohort of patients undergoing an induction of labor. Here, an 11 minute and 30 second counseling video was created to counsel patients on the finer intricacies of an induction of labor. Patients were randomized to two groups: verbal counseling and video + verbal counseling. Patients were randomized just prior to beginning their induction of labor. After receiving verbal counseling or verbal and video counseling, patients completed a survey analyzing their awareness of the counseling process.

DETAILED DESCRIPTION:
This is a Randomized Control Trial where English speaking patients undergoing and induction of labor at the University of Louisville hospital will be randomly assigned to either receive video counseling and verbal counseling or standard verbal counseling alone over the course of 1 year to obtain the desire number of participants. Participants in the video group will also receive standard verbal counseling provided by the resident. Data collection will be Survey based and with use of a lichert scale. Treatment randomization will be performed using a block randomization approach with block sizes of 10 individuals. Random assignments will be made and these will be placed in numbered envelopes to be opened by the intern resident after patient consent is obtained to participate in the study. Eligible participants will be recruited to the study at the time of presentation for their induction of labor. The intern resident will offer them a brief introduction to the project including risks/ benefits to participation and go over the consent process after they have been roomed in a private labor and delivery room. If agreeable to taking part in the study, participants will be given a consent form with an overview of the project with instructions to sign the consent form if agreeable to participating in the study. The intern resident will verbally consent the patient to participate in the study and discuss the study in detail including risks and benefits of participation. All conversations between the subject and co-investigators will take part in the privacy of the patient's labor and delivery room. There will be a short waiting period between the introduction of the study and the patient signing or declining the consent form. This will allow the patient to read the official consent form and ask any remaining questions. After informed consent is obtained, the consent form will be placed in a binder on labor and delivery, to be uploaded into redcap soon thereafter. This binder will be placed in a locked cabinet and only the research personnel identified on this IRB proposal will have access to this cabinet. Those who are randomized to video counseling will watch the counseling video on a portable iPad. This iPad is used for video interpreting on labor and delivery and is on wheels, which will allow for video counseling in any labor and delivery room at any time. This iPad device will be brought to the room by the intern resident. It has already been provided by the Labor and Delivery unit at the University of Louisville hospital. Those randomized to watch the video will watch this video immediately after obtaining consent to participate in the survey. A member of the research team will not be available during the time the patient is viewing the video. It is 10 minutes long. Its content includes introduction to labor and delivery residents, attendings, and staff as well as induction methods, pain control options, expectations for discharge, and common labor and delivery unit protocols including diet and visitors. The video will only be able to viewed by private link to YouTube. This link will be accessible on the iPad homescreen. The video link is as follows: https://www.youtube.com/watch?v=Lbb6E-4iizI. Paper surveys will then be provided to both groups of patients. Surveys will be completed at the exact same time for both groups when official hospital consent is obtained by the resident for cesarean section, vaginal delivery, and blood transfusion. This traditionally occurs after patients have received standard verbal counseling concerning their induction of labor.Those randomized to video counseling will complete the exact survey after completion of the induction of labor video and at the time of official hospital consent. This will ensure both groups of patients are completing the paper survey at the exact same time. Completed surveys and consents will be placed in a binder on labor and delivery in a locked cabinet. The difference in mean cumulative Lichert scores (primary outcome) between the counseling groups will be assessed using the two-sample t-test. Descriptive statistics (sample proportions, mean, standard deviation, etc) will be computed for demographic variables, and comparison between randomization groups will be carried out by chi-squared, Fisher exact, and two-sample t-tests. Linear regression may be used to measure the relationship between demographic variables and counseling experience (primary outcome). Transformations or non-parametrics tests may be used to account for non-normality in response variables. Differences in individual Lichert questions between treatment group may also be run using the t-test or non-parametric Mann-Whitney test. An R Statistical Software will be utilized.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an induction of labor who read, understand, and speak English.
* Patients undergoing an induction of labor who are age 18 and older.
* Any gestational age undergoing an induction of labor.

Exclusion Criteria:

* Patients undergoing an induction of labor who do not read, understand, or speak English.
* Patients undergoing an induction of labor less than age 18.
* Any patients who is admitted under a certified nurse midwife will not be eligible to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Counseling | Up to 1 year
  A patient's awareness of counseling of the process of an induction of labor will be evaluated by lichert scale. A score of 5 (maximum) represents "strongly agree" and a score of 1 (minimum) represents "strongly disagree." Higher scores represent more awareness of the counseling process.

CONTACTS AND LOCATIONS:
Locations (1):
- Univerisity of Louisville Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosaasen N, Mainra R, Kukha-Bryson A, Nhin V, Trivedi P, Shoker A, Wilson J, Padmanabh R, Mansell H. Development of a patient-centered video series to improve education before kidney transplantation. Patient Educ Couns. 2018 Sep;101(9):1624-1629. doi: 10.1016/j.pec.2018.04.014. Epub 2018 Apr 26. PMID 29729857
- [Result] Wilson ME, Krupa A, Hinds RF, Litell JM, Swetz KM, Akhoundi A, Kashyap R, Gajic O, Kashani K. A video to improve patient and surrogate understanding of cardiopulmonary resuscitation choices in the ICU: a randomized controlled trial. Crit Care Med. 2015 Mar;43(3):621-9. doi: 10.1097/CCM.0000000000000749. PMID 25479118
- [Result] Beckmann M, Cooper C, Pocock D. INFORMed choices: facilitating shared decision-making in health care. Aust N Z J Obstet Gynaecol. 2015 Jun;55(3):294-7. doi: 10.1111/ajo.12343. Epub 2015 Jun 5. PMID 26053591
- [Result] Winston K, Grendarova P, Rabi D. Video-based patient decision aids: A scoping review. Patient Educ Couns. 2018 Apr;101(4):558-578. doi: 10.1016/j.pec.2017.10.009. Epub 2017 Oct 18. PMID 29102063
- [Result] Davis SA, Carpenter DM, Blalock SJ, Budenz DL, Lee C, Muir KW, Robin AL, Sleath B. A randomized controlled trial of an online educational video intervention to improve glaucoma eye drop technique. Patient Educ Couns. 2019 May;102(5):937-943. doi: 10.1016/j.pec.2018.12.019. Epub 2018 Dec 18. PMID 30583913
- [Result] Staley SA, Charm SS, Slough LB, Zerden ML, Morse JE. Prenatal Contraceptive Counseling by Video. South Med J. 2019 Jan;112(1):8-13. doi: 10.14423/SMJ.0000000000000913. PMID 30608623
- [Result] Weston J, Hannah M, Downes J. Evaluating the benefits of a patient information video during the informed consent process. Patient Educ Couns. 1997 Mar;30(3):239-45. doi: 10.1016/s0738-3991(96)00968-8. PMID 9104380
- [Result] Greene KA, Wyman AM, Scott LA, Hart S, Hoyte L, Bassaly R. Evaluation of patient preparedness for surgery: a randomized controlled trial. Am J Obstet Gynecol. 2017 Aug;217(2):179.e1-179.e7. doi: 10.1016/j.ajog.2017.04.017. Epub 2017 Apr 18. PMID 28431952
- [Result] Farrell RM, Agatisa PK, Mercer MB, Mitchum AG, Coleridge MB. The use of noninvasive prenatal testing in obstetric care: educational resources, practice patterns, and barriers reported by a national sample of clinicians. Prenat Diagn. 2016 Jun;36(6):499-506. doi: 10.1002/pd.4812. Epub 2016 Apr 7. PMID 26991091
- [Result] Newsom E, Lee E, Rossi A, Dusza S, Nehal K. Modernizing the Mohs Surgery Consultation: Instituting a Video Module for Improved Patient Education and Satisfaction. Dermatol Surg. 2018 Jun;44(6):778-784. doi: 10.1097/DSS.0000000000001473. PMID 29642110
- [Result] Martin JA, Hamilton BE, Sutton PD, Ventura SJ, Mathews TJ, Kirmeyer S, Osterman MJ. Births: final data for 2007. Natl Vital Stat Rep. 2010 Aug 9;58(24):1-85. PMID 21254725
- [Result] Cartwright A. Mothers' experiences of induction. Br Med J. 1977 Sep 17;2(6089):745-9. doi: 10.1136/bmj.2.6089.745. PMID 912282
- [Result] Nuutila M, Halmesmaki E, Hiilesmaa V, Ylikorkala O. Women's anticipations of and experiences with induction of labor. Acta Obstet Gynecol Scand. 1999 Sep;78(8):704-9. PMID 10468063
- [Result] Stewart P. Patients' attitudes to induction and labour. Br Med J. 1977 Sep 17;2(6089):749-52. doi: 10.1136/bmj.2.6089.749. PMID 912283
- [Result] Tong CT, Mackeen AD, Berghella V. The effect of standardized counseling on patient knowledge about induction of labor. J Matern Fetal Neonatal Med. 2012 Dec;25(12):2700-3. doi: 10.3109/14767058.2012.703726. Epub 2012 Jul 13. PMID 22708706